CLINICAL TRIAL: NCT05764460
Title: Social Cognition and Language in Patients With Gliomas: Putting Feelings Into Words
Brief Title: Social Cognition and Language in Patients With Gliomas
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 11351
Record Dates: First submitted 2023-01-25; First posted 2023-03-10 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Glioma, Malignant; Cognitive Dysfunction
MeSH Terms: conditions — Glioma; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Neuropsychological tests — Neuropsychological tests for general cognition, social cognition and language.

SUMMARY:
Patients with gliomas often suffer from lower quality of life, and detrimental social interactions after diagnosis. Two cognitive processes are crucial for maintaining healthy social relationships and interacting with others: social cognition and language. Social cognition is the ability to recognize and process mental and emotional states and to react appropriately in social situations. Social cognition and language are separate cognitive functions that can be affected in different ways in patients with brain injury. Also, distinct cognitive measurement instruments are used to assess both processes. However, there appears to be a certain overlap between social cognition and language. Reacting adequately in social situations requires both verbal and non-verbal communication and to communicate feelings, thoughts and intentions, people often use language. That is, verbal communication is part of a symbolic system that makes social interaction possible. Therefore, language abilities seem to be important to social cognition. Research shows that language is frequently impaired in adult patients with gliomas. Importantly, recent evidence suggests that social cognition can also be impaired in this patient group. However, no studies have been conducted into the relationship between social cognition and language in patients with gliomas. Increasing knowledge on the overlap between both functions, more specifically the influence of language difficulties on social cognition, will improve diagnostic accuracy. Eventually, this will lead to better, tailor-made treatments for these problems that negatively affect daily functioning.

Objective: The main research objective is to examine the influence of language impairments on different social cognition processes, i.e., emotion recognition, Theory of Mind (ToM) and affective empathy, in patients with (suspected) gliomas. Secondary objectives are 1) to determine if patients with gliomas show impairments in different aspects of social cognition, i.e. emotion recognition, ToM, empathy and self-awareness; 2) to assess specific language impairments by looking at item-level characteristics of language tasks (e.g., analyses of word properties of fluency tasks, errors during object naming or spontaneous speech), and 3) to determine which tumor characteristics (low- or high-grade, genetic mutation, tumor location) are associated with different aspects of language and social cognition.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected gliomas, i.e. low- or high-grade gliomas.
* Age older than 18 years
* Sufficient command of the Dutch language
* Being able to understand the instructions of the NPA and to mentally and physically sustain/endure the assessment; this will be assessed in a consultation between treating physician (neurosurgeon) and investigator (neuropsychologist).

Exclusion Criteria:

* Serious neurodegenerative or psychiatric conditions (including addiction)
* Serious (other) medical conditions or physical inability hindering patients to come to the hospital
* Patients who need to undergo emergency craniotomy due to progression of disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a radiologically suspected glioma, referred for surgery (resection or biopt) in the UMCG, department of Neurosurgery, are eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Impairments in emotion recognition | 10 minutes
  FEEST
Impairments in Theory of Mind | 10 minutes
  Cartoons
Impairments in social insight | 10 minutes
  Faux Pas
Impairments in phonology, semantics, syntaxis | 10 minutes (total NPA approximately 3 hours)
  Screeling
Impairments in naming | 5 minutes (total NPA approximately 3 hours)
  Boston Naming Test
Impairments in fluency | 5 minutes (total NPA approximately 3 hours)
  Fluency
Impairments in language comprehension | 5 minutes (total NPA approximately 3 hours)
  SAN

SECONDARY OUTCOMES:
Impairments in memory | 10 minutes (total NPA approximately 3 hours)
  Rivermead Behavioral Memory Test
Impairments in executive functions | 2 minutes (total NPA approximately 3 hours)
  Key Search
Impairments in speed and attention | 5 minutes (total NPA approximately 3 hours)
  Trail Making Test
Impairments in structured spontaneous language | 5 minutes (total NPO approximately 3 hours)
  Cookie Theft
Impairments in general language | 5 minutes (total NPO approximately 3 hours)
  QUEST-NL
Impairments in unstructured spontaneous language | 5 minutes (total NPO approximately 3 hours)
  Story telling
Empathy | Approximately 3 minutes
  Questionnaire filled in by patient and proxy: IRI
Social abilities | Approximately 3 minutes
  Questionnaire filled in by patient and proxy: DEX
Relationship quality | Approximately 4 minutes
  Questionnaire filled in by patient and proxy: CSI